CLINICAL TRIAL: NCT04539444
Title: A Study Evaluated Efficacy and Safety of CD19/22 Chimeric Antigen Receptor T Cells Combined With PD-1 Inhibitor in Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: A Study of CD19/22 CART Cells Combined With PD-1 Inhibitor in Relapsed/Refractory B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCPD-1 in lymphoma
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-08

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
Keywords: Chimeric antigen receptor T cells; Relapsed or refractory B cells non-Hodgkin's lymphoma; PD-1 inhibitor
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — tislelizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/22 CART cells combined with PD-1 inhibitors (Experimental): Patients will receive PD-1 inhibitor on the first day after CART cell infusion
  Interventions: Biological: CD19/22 CART; Drug: Tislelizumab

INTERVENTIONS:
Biological: CD19/22 CART — CD19/22 CART cells are administrated in a 3-day split-dose regimen at dose of 0.5- 2×10*107 CART cells per kilogram of body weight.
Drug: Tislelizumab — Patients will receive Tislelizumab 200mg/dose every 3 weeks.
  Other Names: PD-1 inhibitor

SUMMARY:
This is a single center, non-randomized, open-label, phase 2 study to evaluate the efficacy and safety of CD19/22 CART cells combined with PD-1 Inhibitor in relapsed/refractory B Cell Lymphoma.

DETAILED DESCRIPTION:
Though response rates have greatly improved with the development of Chimeric antigen receptor T cells (CART) therapy in refractory/relapsed B cell non-Hodgkin's lymphoma (R/R B-NHL), the response can't usually last long and relapse occurs in a large proportion of patients who receive CART cells infusion. The main reasons of relapse might be tumor antigen loss and a lack of CART cell persistence. Currently, preclinical studies have shown that there is a synergistic effect between CAR-T cell therapy and anti-PD1 pathway, and it did have efficacy in clinic. In parallel, the combined use of CART-19 and CART-22 cells has a better potential to reduce antigen escape and increase anti-tumor activity. Therefore, the combination of CD19/22 CART and PD-1 inhibitor is one of the ways to improve the therapeutic effect of CART cells. This study was conducted to explore the efficacy and safety of CD19/22 CART cells in R/R B-NHL.

ELIGIBILITY:
Inclusion Criteria:

1. R/R B-NHL with measurable (≧1.5cm) lesions confirmed by pathological immunohistochemistry or flow cytometry ( meeting any of the following conditions):

   A.The lesion shrinkage <50% or disease progression after 4 courses of standard first-line treatment or 2 courses of two-line treatment (primary refractory disease) B. Progress disease as the best response after hematopoietic stem cell transplantation C.Progress disease or stable disease as the best response to most recent therapy regimen
2. Age ≥ 18 years
3. The Eastern Cooperative Oncoloy Group (ECOG) physical condition score ≤ 2 points
4. The main organ functions need to meet the following conditions:

   A.Left ventricular ejection fraction ≥50% B.Creatinine ≤132umol/l or creatinine clearance ≥60 ml/min C.ALT and AST≤2 upper limitation of normal D.SpO2 > 90%
5. Results of pregnant test should be negative, and agree to conception control during treatment and 1 year after CAR-T infusion
6. Expected survival exceeds 3 months
7. Written informed consent could be acquired

Exclusion Criteria:

1. Immunosuppressant medications or steroids was used within 2 weeks before cell collection, or need to use steroids or immunosuppressant medications more than two years
2. Uncontrolled bacteria, fungi, viruses, mycoplasma or other types of infection
3. Active hepatitis B or hepatitis C infection
4. HIV infection
5. Severe acute or chronic graft-versus-host disease (GVHD)
6. Participated in any other drug research clinical trials within 30 days before enrollment
7. Prior CART cells therapy within 3 months before enrollment
8. Prior allogeneic hematopoietic stem cell transplantation within 6 months before enrollment
9. Have contraindications to the PD-1 inhibitors
10. Uncontrolled other tumor
11. Women in pregnancy,lactation or planning to become pregnant
12. The researcher considers inappropriate to participate in this research

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 1 year
  Number of patients who achieved response (complete response and partial response ) after treatment of CD19/22 CART combined with PD-1 inhibitor. Response will be assessed using the Lugano criteria.
Progression-free survival(PFS) | 1 year
  PFS will be assessed from the first CART cell infusion to progression,death or last follow-up.

SECONDARY OUTCOMES:
Complete relapse rate(CR) | 1 year
  Number of patients who achieved complete response after treatment by CD19/22 CART combined with PD-1 inhibitor.
Duration of overall response (DOR) | 1 year
  Duration of overall response will be assessed from the first CAR-T cell infusion to progression,death or last follow-up.
Overall survival(OS) | 1 year
  OS will be assessed from the first CART cell infusion to death or last follow-up.
Incidence of treatment-related adverse events | 1 year
  The incidence rate of adverse events from the first day of preconditioning chemotherapy to 1 year after CART cells infusion

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D., Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China